CLINICAL TRIAL: NCT03063736
Title: Entolimod, an Adjuvant for Vaccine Augmentation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Thomas R. Kosten, MD, Waggoner Chair and Professor of Psychiatry, Neuroscience, Pharmacology, Immunology & Pathology Director, Dan Duncan Institute for Clinical and Translational Research, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-39354
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — CBLB502; Diphtheria-Tetanus Vaccine; Tetanus Toxoid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Td vaccine with entolimod (Experimental): Td vaccine (4 ug) + Entolimod (1 ug) (n=25)
  Interventions: Drug: Entolimod; Biological: Td Vaccine
- Td vaccine only (Placebo Comparator): Td vaccine (4 ug) (n=15)
  Interventions: Biological: Td Vaccine

INTERVENTIONS:
Drug: Entolimod — The objective is to compare adverse events and anti-tetanus (TT) antibody levels between patients getting entolimod vs no entolimod combined with tetanus-diphtheria (Td) vaccine. This clinical trial in 40 normal health subjects compares a single dose of 4 ug Td (2 ug of TT and 2 ug of diphtheria toxoid + 3000 ug of alum) with or without entolimod (1μg).
  Other Names: CBLB502
  Arms: Td vaccine with entolimod
Biological: Td Vaccine — The objective is to compare adverse events and anti-tetanus (TT) antibody levels between patients getting entolimod vs no entolimod combined with tetanus-diphtheria (Td) vaccine. This clinical trial in 40 normal health subjects compares a single dose of 4 ug Td (2 ug of TT and 2 ug of diphtheria toxoid + 3000 ug of alum) with or without entolimod (1μg).
  Other Names: Tetanus and Diphtheria Toxoids Adsorbed

SUMMARY:
The primary objective of this pilot study to evaluate the safety of low dose Entolimod in normal, healthy, non-patient normals. This clinical trial in 40 normal humans compares a single dose of 4 ug Td (2 ug of TT and 2 ug of diphtheria toxoid + 3000 ug of alum with or without entolimod. Subjects will be randomized to: Td alone (n=15) and Td+ entolimod (n=25). The investigators expect that Td + entolimod will double the anti-TT and anti-diphtheria AB levels over Td alone.

DETAILED DESCRIPTION:
This is a single-blind (participants are blinded), pilot study with no therapeutic or diagnostic intent and limited drug exposure. The study will be conducted at Baylor College of Medicine in normal, healthy, and non-drug using male volunteers who have not received the Td vaccination in the past 5 years.

The purpose of this study is to evaluate the safety and surrogate efficacy of low dose entolimod in normal, healthy, non-patient subjects by comparing anti-tetanus (TT) antibody levels between patients getting entolimod vs no entolimod combined with tetanus-diphtheria (Td) vaccine. Subjects will be randomly assigned to one of two arms in a 3:5 ratio (for every 8 subjects, 3 will be randomly assigned to the control group and 5 to the treatment group) to receive a single dose of:

Arm 1: Td (4 ug) (n=15), Arm 2: Td (4 ug) + Entolimod (1 ug) (n=25)

We propose to give the normal dose of Td given routinely to humans (i.e. TT at 2μg and diphtheria toxoid at 2 ug) for a total protein dose of 4 ug. The proposed dose of entolimod at 1 ug is 30-40 times lesser than that previously given safely to humans. We expect that Td + entolimod will double the anti-tetanus toxoid antibody (anti-TT AB) and anti-diphtheria AB levels over Td alone. We predict that this low dosing of entolimod (1μg) produces no difference in adverse effects from giving Td vaccine alone and that any adverse events will be no different than what is typical as reported in the Physicians' Desk Reference for Td vaccine in humans.

For purposes of this trial, study population age cut-off will be 40 years of age. The reason for this cut-off is that the body produces higher antibody levels in response to vaccines in younger age groups compared to older groups. Further, this study is restricted to males only as a safety measure so that women of child-bearing age are not exposed to entolimod, which has not been given to women of childbearing potential.

We consider our strategy adequate for human safety for several reasons related to risks for this new combination of an existing vaccine and new adjuvant. First, our proposed Td-Entolimod starting dose is the usual approved clinical dose of Td (4 μg containing 2 ug TT + 2 ug diphtheria toxoid). Second, the proposed dose for the adjuvant entolimod (1 μg) is supported by both animal toxicology studies and human safety/PK/PD studies cross-referenced from IND 100480. The results of these safety studies, which have given humans up to 30 μg and animals up to 100μg, strongly support that entolimod at 1μg is a safe human dose. The other adjuvant is aluminum phosphate, which is contained within the standard Td vaccine in humans. Third, further support for safety comes from the recent recommendations to boost pregnant women with Td at each pregnancy regardless whether or not they have recently received a Td shot. This recommendation of acceptable enough safety for ACIP to recommend it for pregnant women, supports that this study's single dosing with Td even at less than a 5 year interval would be relatively low risk. Fourth, other FDA approved conjugate vaccines using TT have contained 8 to 10 times greater doses of TT than in our planned dose. Fifth, we will have a randomization of 25 subjects to the Td-Entolimod combination vaccine, which will provide sufficient numbers of subjects to detect common adverse events such as fever and local site reactions in more than one human subject in our vaccinated group compared to the Td alone control group. Local injection site and systemic inflammatory changes also will be monitored in planned clinical study trials with later TT conjugate anti-addiction vaccines.

The close monitoring of objective and subjective drug effects by direct observation, blood work (CBC and Comprehensive Metabolic Panel), weekly telephone check-ins over a 6 week period from point of vaccination to close-out visit to monitor for potential adverse reactions, and a close-out physical will allow objective evaluation of the effects of the vaccines in these normal subjects. We will also have post treatment follow up period with monthly telephone visits up to 1 year from vaccination to further monitor for adverse reactions.

At 6-weeks post-vaccination, we will analyze level of anti-TT AB and anti-diphtheria AB and compare both study arms compared to baseline AB levels to determine the immune potentiating capability of entolimod. In addition to not expecting any difference in adverse events (AE) from giving Td alone compared to those AE listed in the Physicians' Desk Reference for Td in normals, we also expect the AB levels at 6 weeks post vaccination and the ratio of 6-week to baseline AB levels from Td+entolimod (n=25) to be at least double the levels from Td alone (n=15).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-patient normal males between 18 and 40 years of age
2. No baseline anti-TT AB (tetanus toxoid antibody) levels greater than 5 µg/ml
3. Able to read/write/understand English and provide signed written informed consent prior to any study specific procedures.

Exclusion Criteria:

1. Inability to read/write English
2. Inability to provide written informed consent.
3. Any major cardiovascular, renal, endocrine, immunological (including positive test result for human immunodeficiency virus types 1 or 2 antibodies) or hepatic disorder (including positive test result for hepatitis B, hepatitis C virus antibodies, or liver function tests (LFT's)(SGOT, SGPT) that are 20% greater than normal levels or history of severe alcohol use disorder (defined as a score of 5 of greater on the MINI, based on DSM criteria).
4. Medical contraindication to treatment with vaccine as indicated by a history of autoimmune disease, immune deficiency, or hypersensitivity to other vaccines. Specific disorders include a prior Arthus-type hypersensitivity reaction to tetanus vaccine or any of its components, prior Guillain-Barre Syndrome, Ongoing active infection of any kind with clinical signs of febrile illness (temperature >99.5ºF).
5. Use of psychoactive or hepatotoxic medications or medications that might interact with the tetanus toxoid based vaccine including steroids within 30 days of screening, immunosuppressive or immunostimulant therapy.
6. Received other vaccines, including flu vaccine, within 30 days prior to screening or Tetanus vaccine within 5 years of this study (Advisory Committee on Immunization Practices (ACIP) guidelines.
7. Blood or blood products given in the 3 months prior to vaccination.
8. Participation in another investigational pharmaceutical trial within 30 days prior to screening.
9. Greater than Grade 1 abnormality in baseline safety labs (e.g, CBC and CMP), as defined using the FDA Guidance Document entitled "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials"
10. Greater than Grade 1 abnormality in baseline vital signs
11. Women, as a standard safety measure, will be excluded from the study due to childbearing potential and to minimize the effects of differences in hormonal levels during the menstrual cycle and of sex differences in antibody titer responses to vaccines. Furthermore, our sample size is too small to control for these effects in women.
12. Other concerns that in the PI's judgment will be a potential safety issue for the subject including cognitive impairment that precludes the ability to provide informed consent, and individuals with behavioral issues evidenced during screening or through the course of the trial that are disruptive and/or pose a safety concern to self or other subjects.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse events associated with entolimod augmentation. | 6 weeks
  The proposed dose of entolimod used in our study is 30-40 times lesser than that previously given safely to humans. Although our pre-clinical data suggest that these very low levels of entolimod efficiently enhances the antibody levels to TT vaccine in rodents, the safety and success rate at these low doses of entolimod to enhance anti-TT AB in humans requires examination.

SECONDARY OUTCOMES:
Antibody titer comparison with entolimod augmentation of Td vaccine | 6 weeks
  This study will analyze level of anti-TT AB and anti-diphtheria AB and compare both study arms at 6 weeks post vaccination to baseline AB levels to determine the immune potentiating capability of entolimod. We expect the AB levels at 6 weeks post vaccination and the ratio of 6-week to baseline AB levels from Td+entolimod (n=25) to be at least double the levels from Td alone (n=15).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kosten, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krivokrysenko VI, Toshkov IA, Gleiberman AS, Krasnov P, Shyshynova I, Bespalov I, Maitra RK, Narizhneva NV, Singh VK, Whitnall MH, Purmal AA, Shakhov AN, Gudkov AV, Feinstein E. The Toll-Like Receptor 5 Agonist Entolimod Mitigates Lethal Acute Radiation Syndrome in Non-Human Primates. PLoS One. 2015 Sep 14;10(9):e0135388. doi: 10.1371/journal.pone.0135388. eCollection 2015. PMID 26367124
- [Background] Krivokrysenko VI, Shakhov AN, Singh VK, Bone F, Kononov Y, Shyshynova I, Cheney A, Maitra RK, Purmal A, Whitnall MH, Gudkov AV, Feinstein E. Identification of granulocyte colony-stimulating factor and interleukin-6 as candidate biomarkers of CBLB502 efficacy as a medical radiation countermeasure. J Pharmacol Exp Ther. 2012 Nov;343(2):497-508. doi: 10.1124/jpet.112.196071. Epub 2012 Jul 26. PMID 22837010
- [Background] Leigh ND, Bian G, Ding X, Liu H, Aygun-Sunar S, Burdelya LG, Gudkov AV, Cao X. A flagellin-derived toll-like receptor 5 agonist stimulates cytotoxic lymphocyte-mediated tumor immunity. PLoS One. 2014 Jan 14;9(1):e85587. doi: 10.1371/journal.pone.0085587. eCollection 2014. PMID 24454895
- [Background] Howell BA, Siler SQ, Shoda LK, Yang Y, Woodhead JL, Watkins PB. A mechanistic model of drug-induced liver injury AIDS the interpretation of elevated liver transaminase levels in a phase I clinical trial. CPT Pharmacometrics Syst Pharmacol. 2014 Feb 5;3(2):e98. doi: 10.1038/psp.2013.74. PMID 24500662
- [Background] Danilova E, Shiryayev A, Kristoffersen EK, Sjursen H. Attenuated immune response to tetanus toxoid in young healthy men protected against tetanus. Vaccine. 2005 Oct 10;23(42):4980-3. doi: 10.1016/j.vaccine.2005.05.028. PMID 15985319